CLINICAL TRIAL: NCT05255081
Title: A Prospective Single-blind Randomised Controlled Trial Evaluating Clinical Effects of a Novel Spray-Type Bio-absorbable Adhesion Barrier System (AdSpray™) in Paediatric Patients Requiring Laparotomy
Brief Title: Evaluating Clinical Effects of a Spray-Type Bio-absorbable Adhesion Barrier System in Paediatric Patients
Acronym: PEARL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PEARLTrial
Record Dates: First submitted 2022-02-04; First posted 2022-02-24 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2023-05

CONDITIONS: Surgical Adhesions
Keywords: Paediatric surgery; surgical adhesions; medical device; biodegradable anti-adhesive agent
MeSH Terms: conditions — Tissue Adhesions

STUDY DESIGN:
Intervention Model Description: Eligible subjects will be identified, and parents will be approached for patient recruitment. Once consent to participation is signed, the patients will be randomised into either treatment group (AdSpray™) or placebo-controlled group in 1:1 ratio using simple randomization. The adhesion-assessment team will be blinded to the group allocated. The spray will be prepared according to the group allocated by a dedicated scrub nurse. For treatment group, AdSpray™ will be instilled into the drug chamber; for placebo group, saline will be instilled instead.
Who Masked: Participant, Outcomes Assessor
Masking Description: After completion of necessary operative procedures in the primary operation, barrier agent (AdSpray™or Placebo) will be sprayed to fully cover the organs under the laparotomy incision. At the second-look surgery, laparoscopic video recordings of the area under the laparotomy incision will be made in both groups. For the efficacy evaluation, based on the laparoscopic images of the abdominal cavity at the time of the second-look surgery, the presence, extent, and severity of adhesions will be assessed by the adhesion-assessment team which is independent of the study. The independent adhesion-assessment team will assess the extent and severity of adhesions under the laparotomy incision on a 4-grade scale.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Arm (Experimental): Application of AdSpray™ over all organs under the laparotomy incision at the end of operation
  Interventions: Device: Adspray
- Control Arm (Placebo Comparator): Spray with saline would be applied to organs under incision
  Interventions: Procedure: Placebo-control

INTERVENTIONS:
Device: Adspray — Application of AdSpray™ over all organs under the laparotomy incision at the end of operation
  Arms: Treatment Arm
Procedure: Placebo-control — Spray with saline would be applied to organs under incision
  Arms: Control Arm

SUMMARY:
This is a prospective randomized single-blind study where a placebo group served the control, to confirm the efficacy and safety of AdSpray™ as an inhibitory effect of postoperative adhesion formation in paediatric patients who underwent laparotomy with stoma.

DETAILED DESCRIPTION:
Postoperative adhesions are fibrovascular bands connecting the parietal peritoneum to the visceral peritoneum of intra-abdominal organs, or connecting intra-abdominal organs to one another, which developed unavoidably following virtually all body cavity surgeries. Adhesions affect up to 80-93% of patients following abdominal surgery. Being the leading cause of postoperative small bowel obstruction, it could potentially cause other enormous clinical problems including difficulty in subsequent operations, infertility, and chronic pain. The incidence of adhesion-related morbidity is estimated to be 2.2% to 19.5% in the pediatric population, among which large proportion of patients required subsequent surgical intervention. A variety of techniques and products (e.g. bioresorbable physical barrier agents, pharmacological adjuncts, etc) have been advocated for preventing postoperative adhesion formation. However, to date, no single treatment is proven to be effective and adhesions still remain a significant, unresolved postoperative complication both in adults and paediatric populations.

To reduce postoperative adhesions, Terumo Corporation (Tokyo, Japan) has developed an adhesion barrier system (AdSpray™; Terumo Corporation, Tokyo, Japan) which is easy to use at the treatment site in various surgical procedures. Its ability of adhesion prevention had been demonstrated in porcine model study. Cezar et al and Suto et al subsequently published two human prospective randomized controlled trials on the use of this barrier system in adult patients undergoing gynaecological and gastrointestinal operations, which confirmed its safety and efficacy. However, to date, studies on the use of anti-adhesion agents in children are scarce and there is no study on this novel barrier system (AdSpray™) in children. In view of this, we plan to conduct a prospective randomized single-blind study where a placebo group served the control, to confirm the efficacy and safety of AdSpray™ as an inhibitory effect of postoperative adhesion formation in paediatric patients who underwent laparotomy with stoma.

B. Study objective To investigate the effect of a novel spray-type, novel dextrin hydrogel adhesion barrier (AdSpray™; Terumo Corporation, Tokyo, Japan) on postsurgical adhesions.

C. Study design and methods This is a prospective, single center, single-blinded randomized controlled trial using a parallel arm design and placebo group as the control. Patient enrollment will start in March 2022 and expected to end in 2023.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring laparotomy and staged operation with closure of stoma as second operation e.g. Necrotising Enterocolitis, Anorectal malformation, Hirschsprung's disease, etc.

Exclusion Criteria:

* A history of hypersensitivity to substances derived from corn starch
* A history of surgery in the abdominal cavity or pelvic cavity accompanied by a laparotomy scar
* Patients with peritonitis
* Laparoscopic assessment of adhesions may not be performed safely at the second-look surgery.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Incidence of adhesion | 6 months
  The number of participants developed adhesion during the study period at the second operation assessment
Extent of adhesion | 6 months
  Extent of adhesion is classified into 4 grade: Grade 0 - none, Grade 1 - adhesion less than 1/3 the length of incision, Grade 2 - adhesions between 1/3 and <2/3 the length of the incision, Grade 3 - Adhesion great or equal than 2/3 the length of the incision
Severity of adhesion | 6 months
  Severity of adhesion is classified into 4 grade: Grade 0 - none, Grade 1 - film-like with no neovascularisation, Grade 2 - moderately thick with partial neovascularisation, Grade 3 - thick, solid adhesion with neovascularisation

SECONDARY OUTCOMES:
Adverse events | 6 months
  Intestinal obstruction, abscess, peritonitis, surgical wound infection, malfunction of device, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Chi Heng Fung, MBBS, Principal Investigator — The University of Hong Kong
Locations (1):
- Department of Surgery, University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thakur M, Rambhatla A, Qadri F, Chatzicharalampous C, Awonuga M, Saed G, Diamond MP, Awonuga AO. Is There a Genetic Predisposition to Postoperative Adhesion Development? Reprod Sci. 2021 Aug;28(8):2076-2086. doi: 10.1007/s43032-020-00356-7. Epub 2020 Oct 22. PMID 33090376
- [Background] Foster DS, Marshall CD, Gulati GS, Chinta MS, Nguyen A, Salhotra A, Jones RE, Burcham A, Lerbs T, Cui L, King ME, Titan AL, Ransom RC, Manjunath A, Hu MS, Blackshear CP, Mascharak S, Moore AL, Norton JA, Kin CJ, Shelton AA, Januszyk M, Gurtner GC, Wernig G, Longaker MT. Elucidating the fundamental fibrotic processes driving abdominal adhesion formation. Nat Commun. 2020 Aug 13;11(1):4061. doi: 10.1038/s41467-020-17883-1. PMID 32792541
- [Background] Lakshminarayanan B, Hughes-Thomas AO, Grant HW. Epidemiology of adhesions in infants and children following open surgery. Semin Pediatr Surg. 2014 Dec;23(6):344-8. doi: 10.1053/j.sempedsurg.2014.06.005. Epub 2014 Jun 4. PMID 25459439
- [Background] Nguyen ATM, Holland AJA. Paediatric adhesive bowel obstruction: a systematic review. Pediatr Surg Int. 2021 Jun;37(6):755-763. doi: 10.1007/s00383-021-04867-5. Epub 2021 Apr 19. PMID 33876300
- [Background] Inoue M, Uchida K, Otake K, Nagano Y, Ide S, Hashimoto K, Matsushita K, Koike Y, Mohri Y, Kusunoki M. Efficacy of Seprafilm for preventing adhesive bowel obstruction and cost-benefit analysis in pediatric patients undergoing laparotomy. J Pediatr Surg. 2013 Jul;48(7):1528-34. doi: 10.1016/j.jpedsurg.2013.01.028. PMID 23895967
- [Background] Kai M, Maeda K, Tasaki M, Kira S, Nakamura S, Chino N, Hagiwara H, Nishida H, Kawanishi T. Evaluation of a Spray-type, Novel Dextrin Hydrogel Adhesion Barrier Under Laparoscopic Conditions in a Porcine Uterine Horn Adhesion Model. J Minim Invasive Gynecol. 2018 Mar-Apr;25(3):447-454. doi: 10.1016/j.jmig.2017.09.023. Epub 2017 Oct 10. PMID 29030291
- [Background] Suto T, Watanabe M, Endo T, Komori K, Ohue M, Kanemitsu Y, Itou M, Takii Y, Yatsuoka T, Shiozawa M, Kinugasa T, Ueno H, Takayama T, Masaki T, Masuko H, Horie H, Inomata M. The Primary Result of Prospective Randomized Multicenter Trial of New Spray-Type Bio-absorbable Adhesion Barrier System (TCD-11091) Against Postoperative Adhesion Formation. J Gastrointest Surg. 2017 Oct;21(10):1683-1691. doi: 10.1007/s11605-017-3503-1. Epub 2017 Jul 25. PMID 28744742
- [Background] Cezar C, Korell M, Tchartchian G, Ziegler N, Senshu K, Herrmann A, Larbig A, De Wilde RL. How to avoid risks for patients in minimal-access trials: Avoiding complications in clinical first-in-human studies by example of the ADBEE study. Best Pract Res Clin Obstet Gynaecol. 2016 Aug;35:84-96. doi: 10.1016/j.bpobgyn.2015.11.004. Epub 2015 Nov 14. PMID 26707194